CLINICAL TRIAL: NCT00249795
Title: A Parallel Randomized Controlled Evaluation of Clopidogrel Plus Aspirin, With Factorial Evaluation of Irbesartan, for the Prevention of Vascular Events, in Patients With Atrial Fibrillation
Brief Title: Atrial Fibrillation Clopidogrel Trial With Irbesartan for Prevention of Vascular Events (ACTIVE I)
Acronym: ACTIVE I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: ICD Study Director, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EFC4912 I; Clopidogrel (SR25990)
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-09

CONDITIONS: Atrial Fibrillation; Cardiovascular Disease
Keywords: Atrial fibrillation; Cardiovascular disease; angiotensin II blocker
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irbesartan (Experimental): 150 mg for 2 weeks, then up-titrated to 300 mg up to final follow-up visit
  Interventions: Drug: Irbesartan
- Placebo (Placebo Comparator): Matching placebo up to final follow-up visit
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Irbesartan — oral administration (tablets) once daily
  Other Names: Aprovel®
  Arms: Irbesartan
Drug: placebo — oral administration (tablets) once daily
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine if Irbesartan compared to Placebo would reduce the risk of vascular events such as heart attack, stroke, non-cerebral thromboembolic event and death in patients with Atrial Fibrillation (AF) and with at least one major risk of vascular events.

DETAILED DESCRIPTION:
ACTIVE I was one of the 3 separate but related trials of the ACTIVE program conducted in AF patients at risk of vascular events.

Patients were enrolled first into one of the 2 parallel trials of the ACTIVE program evaluating Clopidogrel:

* ACTIVE A comparing clopidogrel + acetylsalicylic acid (ASA) and ASA alone
* ACTIVE W comparing clopidogrel + ASA and oral anticoagulant (OAC).

Then those satisfying additional criteria related to blood pressure and angiotensin receptor blocking agents were re-randomized in the two ACTIVE I arms according to a separate randomization list.

ELIGIBILITY:
Inclusion Criteria:

Should fulfill the eligibility criteria for ACTIVE A or ACTIVE W trial and:

* have a systolic blood pressure of at least 110 mmHg
* not already receiving an angiotensin receptor blocking agent, unless they are willing and able to be changed to another antihypertensive agent
* no previous intolerance to angiotensin receptor blocking agents
* no proven indication for angiotensin receptor blocking agents, unless an Angiotensin Converting Enzyme (ACE) inhibitor can be substituted

Exclusion Criteria:

Patients will be excluded from ACTIVE study if any of the following are present:

* requirement for clopidogrel (such as recent coronary stent procedure)
* requirement for oral anticoagulant (such as prosthetic mechanical heart valve)
* prior intolerance to acetylsalicyclic acid (ASA) or clopidogrel
* documented peptic ulcer disease within the previous 6 months
* prior intracerebral hemorrhage
* significant thrombocytopenia (platelet count <50 x 10(9)/L)
* psychosocial reason making study participation impractical
* geographic reason making study participation impractical
* ongoing alcohol abuse
* mitral stenosis
* pregnant or nursing woman or woman of child bearing potential and not on effective birth control for at least one month prior to start of study or not willing to continue on birth control for duration of study
* severe comorbid condition such that the patient is not expected to survive 6 months
* patient currently receiving an investigational pharmacologic agent
* requirement for chronic (> 3 months) non-cyclooxygenase-2 (non-COX-2) inhibitor nonsteroidal anti-inflammatory drug (NSAID) therapy unless willing enrolled in ACTIVE A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9016 (Actual)
Dates: Start 2003-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salim YUSUF, Prof., Study Chair — Hamilton Health Sciences Corporation
Locations (30):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Derived] ACTIVE I Investigators; Yusuf S, Healey JS, Pogue J, Chrolavicius S, Flather M, Hart RG, Hohnloser SH, Joyner CD, Pfeffer MA, Connolly SJ. Irbesartan in patients with atrial fibrillation. N Engl J Med. 2011 Mar 10;364(10):928-38. doi: 10.1056/NEJMoa1008816. PMID 21388310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in 567 centers in 33 countries. They were initially to be followed until November 2008. After a blinded reassessment of the event rate in May 2008, the planned follow-up end date was postponed and was actually completed on August 2009 corresponding to an actual median follow-up of 4.5 years.
Groups:
- Irbesartan: 150 mg for 2 weeks, then uptitrated to 300 mg up to final follow-up visit
Period: Overall Study
Arm/Group | Irbesartan | Placebo
Started | 4518 (randomized patients: patients remained in the study whether treated or not until planned study end) | 4498 (randomized patients: patients remained in the study whether treated or not until planned study end)
Completed | 3124 (started and completed study drug) | 3108 (started and completed study drug)
Not Completed | 1394 | 1390
Not completed — Not treated | 16 | 14
Not completed — Symptomatic hypotension | 127 | 64
Not completed — Other Serious Adverse Event | 84 | 93
Not completed — Qualifying condition not present | 26 | 29
Not completed — Withdrawal by Subject | 678 | 742
Not completed — Thromboembolic / outcome event | 39 | 45
Not completed — Oral anticoagulant required | 2 | 0
Not completed — Minor bleeding (e.g.,bruising,epistaxis) | 7 | 3
Not completed — Non-compliance | 71 | 69
Not completed — Study drug intolerance | 3 | 3
Not completed — Other adverse events (non-serious) | 188 | 159
Not completed — Physician withdrew consent | 71 | 63
Not completed — Surgery / procedure | 4 | 5
Not completed — Angiotensin II receptor blocker required | 35 | 58
Not completed — Lightheadedness / dizziness | 15 | 11
Not completed — Hypotension (non-symptomatic) | 5 | 5
Not completed — Other contraindicated medication | 1 | 1
Not completed — Event related to cardiac condition | 17 | 16
Not completed — Patient not wish to continue after May08 | 4 | 6
Not completed — Site not agree to continue after May08 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Missing | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irbesartan | Placebo | Total
Number analyzed (Participants) | 4518 | 4498 | 9016
Age Continuous [Mean (Standard Deviation); unit: years] | 69.5 (9.7) | 69.6 (9.7) | 69.6 (9.7)
Age, Customized [Number; unit: participants]
  18 to <65 years | 1287 | 1255 | 2542
  65 to <75 years | 1684 | 1673 | 3357
  >=75 years | 1547 | 1570 | 3117
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1773 | 1768 | 3541
  Male | 2745 | 2730 | 5475
Congestive heart failure, High blood pressure, Age, Diabetes Stroke 2 (CHADS2) Score [Number; unit: participants] — 7-point, ordinal score determining the risk of stroke from 0 (absence of risk) to 6 (higher risk) depending on the presence or absence of co-morbidities such as history of Congestive heart failure, hypertension, Age, history of Diabetes, previous Stroke.
  participants
    0 | 103 | 96 | 199
    1 | 1687 | 1678 | 3365
    2 | 1516 | 1560 | 3076
    > 2 | 1210 | 1163 | 2373
    Missing | 2 | 1 | 3
Sitting Systolic Blood Pressure [Number; unit: participants]
  <120 mmHg | 509 | 500 | 1009
  >=120 mmHg | 4006 | 3996 | 8002
  Missing | 3 | 2 | 5
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 29.129 (5.614) | 28.867 (5.420) | 28.998 (5.519)
ACTIVE A / ACTIVE W [Number; unit: participants] — Distribution of the patients according to their initial randomization in the ACTIVE program
  participants
    ACTIVE A: clopidogrel + ASA | 1263 | 1231 | 2494
    ACTIVE A: ASA | 1245 | 1259 | 2504
    ACTIVE W: clopidogrel + ASA | 1011 | 959 | 1970
    ACTIVE W: OAC | 999 | 1049 | 2048

OUTCOME MEASURES:

1. Primary Outcome: First Occurence of Any Component of the Composite of Myocardial Infarction, Stroke or Vascular Death as Per Adjudication
Description: The first co-primary event is the first occurence of any component of the following cluster over the duration of follow-up: myocardial infarction (nonfatal or fatal), stroke (nonfatal or fatal) or vascular death - after validation by the Event Adjudication Committee (EAC).
Time Frame: Median follow-up of 4.5 years
Population: The intent-to-treat (ITT) population was used for all analyses. This consisted of all randomized patients irrespective of whether or not the patient actually received study drug or the patient's compliance with the study protocol. All patients were included in the treatment group to which they were originally allocated.
Measure: Number; unit: participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 4518 | 4498
participants
  All components | 963 | 963
  - Myocardial Infarction (fatal or not) | 136 | 123
  - Stroke (fatal or not) | 367 | 407
  - Vascular death | 460 | 433
Statistical Analysis 1: Comparison: Irbesartan vs Placebo; Test type: Superiority or Other; p = 0.8570, Log Rank — The cumulative incidence function of this event was calculated for each treatment group using the non-parametric Kaplan-Meier method and the comparison was performed using a 2-sided Log Rank test at 4.5% level to account for multiplicity; Logrank statistic was stratified on ACTIVE A/W strata; Hazard Ratio (HR) = 0.992, 95% CI 2-sided [0.907 to 1.085] — HR was estimated using a Cox's proportional hazard model stratified on ACTIVE A/W strata with treatment group factor. It provides the relative hazard of any component of the composite event in Irbesartan group versus Placebo group

2. Primary Outcome: First Occurence of Any Component of the Composite of Myocardial Infarction, Stroke, Vascular Death or Hospitalization for Heart Failure as Per Adjudication
Description: The second co-primary event is the first occurence of any component of the following cluster over the duration of follow-up: myocardial infarction (nonfatal or fatal), stroke (nonfatal or fatal), vascular death or hospitalization for heart failure - after validation by the EAC.
Time Frame: Median follow-up of 4.5 years
Population: The intent-to-treat (ITT) population was used for this analysis.
Measure: Number; unit: participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 4518 | 4498
participants
  All components | 1236 | 1291
  - Myocardial Infarction (fatal or not) | 122 | 112
  - Stroke (fatal or not) | 340 | 375
  - Vascular death | 331 | 291
  - Hospitalization for heart failure | 443 | 513
Statistical Analysis 1: Comparison: Irbesartan vs Placebo; Test type: Superiority or Other; p = 0.1200, Log Rank — The cumulative incidence function of this event was calculated for each treatment group using the non-parametric Kaplan-Meier method and the comparison was performed using a 2-sided Log Rank test at 1% level to account for multiplicity; Logrank statistic was stratified on ACTIVE A/W strata; Hazard Ratio (HR) = 0.940, 95% CI 2-sided [0.869 to 1.016] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: First Occurrence of Stroke
Description: The considered event is the first occurrence of stroke (nonfatal or fatal, ischemic, hemorrhagic or of uncertain type) over the duration of follow-up, after validation by the EAC.
Time Frame: Median follow-up of 4.5 years
Population: The intent-to-treat (ITT) population was used for this analysis.
Measure: Number; unit: participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 4518 | 4498
participants | 379 | 411
Statistical Analysis 1: Comparison: Irbesartan vs Placebo; Test type: Superiority or Other; p = 0.2162, Log Rank — The cumulative incidence function of this event was calculated for each treatment group using the non-parametric Kaplan-Meier method and the comparison was performed using a 2-sided Log Rank test at 5% level; Logrank statistic was stratified on ACTIVE A/W strata; Hazard Ratio (HR) = 0.916, 95% CI 2-sided [0.796 to 1.053] — HR was estimated using a Cox's proportional hazard model stratified on ACTIVE A/W strata with treatment group factor. It provides the relative hazard of a stroke in Irbesartan group versus Placebo group

4. Secondary Outcome: Death From Any Cause
Description: The considered event is the death over the duration of the follow-up whatever the cause, cardiovascular or non-cardiovascular.
Time Frame: Median follow-up of 4.5 years
Population: The intent-to-treat (ITT) population was used for the analysis.
Measure: Number; unit: participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 4518 | 4498
participants | 949 | 929
Statistical Analysis 1: Comparison: Irbesartan vs Placebo; Test type: Superiority or Other; p = 0.7590, Log Rank — [p-value comment as in outcome 3, analysis 1]; Logrank statistic was stratified on ACTIVE A/W strata; Hazard Ratio (HR) = 1.014, 95% CI 2-sided [0.927 to 1.110] — HR was estimated using a Cox's proportional hazard model stratified on ACTIVE A/W strata with treatment group factor. It provides the relative hazard of death in Irbesartan group versus Placebo group

5. Secondary Outcome: First Occurrence of Any Heart Failure (HF) Episode
Description: The considered event is the first occurence of any HF episode defined as evidence of signs and symptoms of HF with or without hospitalization over the duration of follow-up, as reported by the investigator (i.e. not validated by the Event Adjudication Committee).
Time Frame: Median follow-up of 4.5 years
Population: The intent-to-treat (ITT) population was used for the analysis.
Measure: Number; unit: participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 4518 | 4498
participants | 699 | 767
Statistical Analysis 1: Comparison: Irbesartan vs Placebo; Test type: Superiority or Other; p = 0.0369, Log Rank — [p-value comment as in outcome 3, analysis 1]; Logrank statistic was stratified on ACTIVE A/W strata; Hazard Ratio (HR) = 0.897, 95% CI 2-sided [0.809 to 0.993] — HR was estimated using a Cox's proportional hazard model stratified on ACTIVE A/W strata with treatment group factor. It provides the relative hazard of HF episodes in Irbesartan group versus Placebo group

6. Secondary Outcome: First Hospitalisation for Heart Failure (HF)
Description: The considered event is the first overnight hospital stay for HF over the duration of the follow-up, after validation by the EAC.
Time Frame: Median follow-up of 4.5 years
Population: The intent-to-treat (ITT) population was used for this analysis.
Measure: Number; unit: participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 4518 | 4498
participants | 482 | 551
Statistical Analysis 1: Comparison: Irbesartan vs Placebo; Test type: Superiority or Other; p = 0.0175, Log Rank — [p-value comment as in outcome 3, analysis 1]; Logrank statistic was stratified on ACTIVE A/W strata; Hazard Ratio (HR) = 0.863, 95% CI 2-sided [0.763 to 0.975] — HR was estimated using a Cox's proportional hazard model stratified on ACTIVE A/W strata with treatment group factor. It provides the relative hazard of hospitalization for Heart Failure in Irbesartan group versus Placebo group

7. Secondary Outcome: First Hospitalisation for Other Cardiovascular (CV) Cause
Description: The considered event is the overnight hospital stay for any CV cause other than Heart Failure over the duration of follow-up, as reported by the investigator (i.e. not validated by the Event Adjudication Committee).
Time Frame: Median follow-up of 4.5 years
Population: The intent-to-treat (ITT) population was used for the analysis.
Measure: Number; unit: participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 4518 | 4498
participants | 1186 | 1174
Statistical Analysis 1: Comparison: Irbesartan vs Placebo; Test type: Superiority or Other; p = 0.8377, Log Rank — [p-value comment as in outcome 3, analysis 1]; Logrank statistic was stratified on ACTIVE A/W strata; Hazard Ratio (HR) = 1.008, 95% CI 2-sided [0.930 to 1.093] — HR was estimated using a Cox's proportional hazard model stratified on ACTIVE A/W strata with treatment group factor. It provides the relative hazard of hospitalization for other CV cause in Irbesartan group versus Placebo group

ADVERSE EVENTS:
Time Frame: From randomization until 14 days after treatment discontinuation or final follow-up visit whichever come first.
Description: The safety analysis was also carried out on the intent-to-treat (ITT) population to allow a benefit/risk assessment within the same study population.
Arm/Group | Irbesartan | Placebo
Serious Adverse Events (participants affected / at risk) | 1409/4518 | 1446/4498
Other Adverse Events (participants affected / at risk) | 3303/4518 | 3277/4498
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irbesartan (N=4518) | Placebo (N=4498)
Pneumonia (Infections and infestations) | 141 | 167
Urinary tract infection (Infections and infestations) | 28 | 26
Bronchitis (Infections and infestations) | 26 | 23
Sepsis (Infections and infestations) | 20 | 28
Gastroenteritis (Infections and infestations) | 19 | 20
Bronchopneumonia (Infections and infestations) | 16 | 18
Cellulitis (Infections and infestations) | 13 | 21
Appendicitis (Infections and infestations) | 10 | 7
Diverticulitis (Infections and infestations) | 10 | 5
Septic shock (Infections and infestations) | 9 | 13
Erysipelas (Infections and infestations) | 9 | 12
Lower respiratory tract infection (Infections and infestations) | 8 | 5
Respiratory tract infection (Infections and infestations) | 6 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 8
Viral infection (Infections and infestations) | 5 | 5
Lung infection (Infections and infestations) | 5 | 2
Urosepsis (Infections and infestations) | 4 | 8
Postoperative wound infection (Infections and infestations) | 4 | 5
Infection (Infections and infestations) | 4 | 2
Haematoma infection (Infections and infestations) | 4 | 0
Lobar pneumonia (Infections and infestations) | 3 | 7
Influenza (Infections and infestations) | 3 | 6
Pyelonephritis (Infections and infestations) | 3 | 6
Wound infection (Infections and infestations) | 3 | 4
Pyelonephritis acute (Infections and infestations) | 3 | 3
Clostridium difficile colitis (Infections and infestations) | 3 | 1
Staphylococcal infection (Infections and infestations) | 3 | 1
Appendicitis perforated (Infections and infestations) | 3 | 0
Clostridial infection (Infections and infestations) | 3 | 0
Tracheobronchitis (Infections and infestations) | 3 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 5
Gangrene (Infections and infestations) | 2 | 3
Herpes zoster (Infections and infestations) | 2 | 3
Post procedural infection (Infections and infestations) | 2 | 3
Bronchiectasis (Infections and infestations) | 2 | 2
Arthritis infective (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 2 | 1
Pulmonary sepsis (Infections and infestations) | 2 | 1
Endocarditis (Infections and infestations) | 2 | 0
Lung infection pseudomonal (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 5
Pulmonary tuberculosis (Infections and infestations) | 1 | 4
Anal abscess (Infections and infestations) | 1 | 2
Cystitis (Infections and infestations) | 1 | 2
Labyrinthitis (Infections and infestations) | 1 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 2
Vestibular neuronitis (Infections and infestations) | 1 | 2
Bacterial pyelonephritis (Infections and infestations) | 1 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 1
Orchitis (Infections and infestations) | 1 | 1
Post procedural sepsis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Anogenital warts (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Encephalitis viral (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Genitourinary tract infection (Infections and infestations) | 1 | 0
Hepatitis e (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Injection site infection (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Peritoneal infection (Infections and infestations) | 1 | 0
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Staphylococcal toxaemia (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Tetanus (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 3
Dengue fever (Infections and infestations) | 0 | 3
Localised infection (Infections and infestations) | 0 | 3
Gallbladder empyema (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 2
Pneumonia primary atypical (Infections and infestations) | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 0 | 1
Appendiceal abscess (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Borrelia infection (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Carbuncle (Infections and infestations) | 0 | 1
Cholangitis suppurative (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Fungal sepsis (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Perinephric abscess (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Splenic abscess (Infections and infestations) | 0 | 1
Thrombophlebitis septic (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Toxic shock syndrome (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 26 | 27
Inguinal hernia (Gastrointestinal disorders) | 20 | 27
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 20 | 15
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 16 | 16
Diarrhoea (Gastrointestinal disorders) | 11 | 7
Gastritis (Gastrointestinal disorders) | 10 | 12
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 | 12
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Colonic polyp (Gastrointestinal disorders) | 8 | 5
Gastritis haemorrhagic (Gastrointestinal disorders) | 7 | 6
Ileus (Gastrointestinal disorders) | 7 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 6 | 10
Gastric ulcer (Gastrointestinal disorders) | 6 | 6
Vomiting (Gastrointestinal disorders) | 6 | 5
Intestinal obstruction (Gastrointestinal disorders) | 5 | 6
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 4 | 8
Pancreatitis (Gastrointestinal disorders) | 4 | 4
Peritonitis (Gastrointestinal disorders) | 4 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 7
Abdominal hernia (Gastrointestinal disorders) | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 5
Retroperitoneal haematoma (Gastrointestinal disorders) | 3 | 4
Umbilical hernia (Gastrointestinal disorders) | 3 | 4
Abdominal strangulated hernia (Gastrointestinal disorders) | 3 | 3
Ascites (Gastrointestinal disorders) | 3 | 1
Diverticulum (Gastrointestinal disorders) | 3 | 1
Food poisoning (Gastrointestinal disorders) | 3 | 1
Rectal polyp (Gastrointestinal disorders) | 3 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 3 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 | 8
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 7
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 4
Colitis ulcerative (Gastrointestinal disorders) | 2 | 3
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 3
Peptic ulcer (Gastrointestinal disorders) | 2 | 3
Duodenal ulcer (Gastrointestinal disorders) | 2 | 2
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 2 | 1
Mechanical ileus (Gastrointestinal disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Volvulus (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 7
Haemorrhoids (Gastrointestinal disorders) | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Melaena (Gastrointestinal disorders) | 1 | 4
Subileus (Gastrointestinal disorders) | 1 | 4
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 2
Duodenitis (Gastrointestinal disorders) | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 2
Gastroduodenitis (Gastrointestinal disorders) | 1 | 2
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 2
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 2
Small intestinal perforation (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric mucosal lesion (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrooesophagitis (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0
Mesenteric occlusion (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Polyp colorectal (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 4
Hiatus hernia (Gastrointestinal disorders) | 0 | 4
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 3
Anal fissure (Gastrointestinal disorders) | 0 | 2
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Anal prolapse (Gastrointestinal disorders) | 0 | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gallstone ileus (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1
Lumbar hernia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 1
Radicular cyst (Gastrointestinal disorders) | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Sigmoiditis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 | 34
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 18
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 15
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 8
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 10
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 8
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 8
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 6
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cystosarcoma phyllodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diaphragm neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymph node cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vascular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 26 | 24
Femur fracture (Injury, poisoning and procedural complications) | 16 | 29
Hip fracture (Injury, poisoning and procedural complications) | 16 | 17
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 14 | 14
Subdural haematoma (Injury, poisoning and procedural complications) | 14 | 11
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 8 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 7 | 7
Ankle fracture (Injury, poisoning and procedural complications) | 6 | 7
Head injury (Injury, poisoning and procedural complications) | 6 | 7
Spinal fracture (Injury, poisoning and procedural complications) | 5 | 9
Overdose (Injury, poisoning and procedural complications) | 5 | 7
Operative haemorrhage (Injury, poisoning and procedural complications) | 5 | 4
Upper limb fracture (Injury, poisoning and procedural complications) | 5 | 3
Facial bones fracture (Injury, poisoning and procedural complications) | 5 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 5 | 2
Drug toxicity (Injury, poisoning and procedural complications) | 5 | 1
Injury (Injury, poisoning and procedural complications) | 4 | 9
Contusion (Injury, poisoning and procedural complications) | 4 | 7
Humerus fracture (Injury, poisoning and procedural complications) | 4 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 3
Concussion (Injury, poisoning and procedural complications) | 4 | 2
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 4 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 4 | 2
Fracture (Injury, poisoning and procedural complications) | 4 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 3 | 4
Anaemia postoperative (Injury, poisoning and procedural complications) | 3 | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 3 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 3 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 4
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 4
Radius fracture (Injury, poisoning and procedural complications) | 2 | 3
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 2
Chest injury (Injury, poisoning and procedural complications) | 2 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 2 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Open fracture (Injury, poisoning and procedural complications) | 2 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 2 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 5
Rib fracture (Injury, poisoning and procedural complications) | 1 | 4
Joint injury (Injury, poisoning and procedural complications) | 1 | 3
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 2
Face injury (Injury, poisoning and procedural complications) | 1 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 1
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Back crushing (Injury, poisoning and procedural complications) | 1 | 0
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 1 | 0
Device failure (Injury, poisoning and procedural complications) | 1 | 0
Dural tear (Injury, poisoning and procedural complications) | 1 | 0
Epiphyseal fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural stroke (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 3
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 2
Accidental poisoning (Injury, poisoning and procedural complications) | 0 | 1
Bladder injury (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Complication of device insertion (Injury, poisoning and procedural complications) | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Pacemaker complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 45 | 40
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 20
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 8
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 4 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal mucosa atrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 58 | 48
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 6
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 9 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 6
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 3
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis enteropathic (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Senile ankylosing vertebral hyperostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Senile osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral wedging (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 35 | 19
Renal failure (Renal and urinary disorders) | 26 | 13
Haematuria (Renal and urinary disorders) | 11 | 11
Renal failure chronic (Renal and urinary disorders) | 7 | 3
Nephrolithiasis (Renal and urinary disorders) | 4 | 5
Haemorrhage urinary tract (Renal and urinary disorders) | 4 | 2
Calculus ureteric (Renal and urinary disorders) | 4 | 1
Urinary retention (Renal and urinary disorders) | 3 | 9
Urethral stenosis (Renal and urinary disorders) | 3 | 5
Renal cyst (Renal and urinary disorders) | 3 | 2
Renal colic (Renal and urinary disorders) | 2 | 3
Calculus urinary (Renal and urinary disorders) | 2 | 2
Urinary bladder polyp (Renal and urinary disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 2
Ureteric stenosis (Renal and urinary disorders) | 1 | 2
Anuria (Renal and urinary disorders) | 1 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Stress urinary incontinence (Renal and urinary disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Bladder stenosis (Renal and urinary disorders) | 0 | 1
Cystitis ulcerative (Renal and urinary disorders) | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Urethral fistula (Renal and urinary disorders) | 0 | 1
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1
Syncope (Nervous system disorders) | 22 | 26
Haemorrhagic stroke (Nervous system disorders) | 13 | 28
Haemorrhage intracranial (Nervous system disorders) | 8 | 13
Dizziness (Nervous system disorders) | 8 | 11
Dementia alzheimer's type (Nervous system disorders) | 5 | 1
Dementia (Nervous system disorders) | 4 | 5
Presyncope (Nervous system disorders) | 4 | 1
Convulsion (Nervous system disorders) | 3 | 10
Polyneuropathy (Nervous system disorders) | 3 | 3
Sciatica (Nervous system disorders) | 3 | 3
Cervical root pain (Nervous system disorders) | 3 | 0
Loss of consciousness (Nervous system disorders) | 3 | 0
Epilepsy (Nervous system disorders) | 2 | 6
Vascular encephalopathy (Nervous system disorders) | 2 | 4
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 2 | 1
Aphasia (Nervous system disorders) | 2 | 0
Vascular dementia (Nervous system disorders) | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 4
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 1 | 3
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 3
Cerebral haemorrhage (Nervous system disorders) | 1 | 2
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1
Dizziness postural (Nervous system disorders) | 1 | 1
Encephalitis (Nervous system disorders) | 1 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 1
Ageusia (Nervous system disorders) | 1 | 0
Anosmia (Nervous system disorders) | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Brachial plexopathy (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Hypokinesia (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Simple partial seizures (Nervous system disorders) | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 2
Intracranial haematoma (Nervous system disorders) | 0 | 2
Paresis (Nervous system disorders) | 0 | 2
Parkinson's disease (Nervous system disorders) | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 2
Anoxic encephalopathy (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral cyst (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1
Mononeuropathy (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 1
Myxoedema coma (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Phantom pain (Nervous system disorders) | 0 | 1
Postictal paralysis (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 29 | 22
Cholecystitis (Hepatobiliary disorders) | 15 | 18
Cholecystitis acute (Hepatobiliary disorders) | 7 | 16
Jaundice (Hepatobiliary disorders) | 4 | 2
Bile duct stone (Hepatobiliary disorders) | 4 | 1
Biliary colic (Hepatobiliary disorders) | 2 | 2
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 4
Cholangitis (Hepatobiliary disorders) | 1 | 3
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Hypotension (Vascular disorders) | 15 | 3
Haemorrhage (Vascular disorders) | 8 | 7
Haematoma (Vascular disorders) | 4 | 6
Hypertension (Vascular disorders) | 4 | 3
Aortic aneurysm (Vascular disorders) | 2 | 8
Bleeding varicose vein (Vascular disorders) | 2 | 2
Thrombophlebitis (Vascular disorders) | 2 | 2
Varicose vein (Vascular disorders) | 2 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 2
Arteriosclerosis (Vascular disorders) | 1 | 2
Arteriosclerosis obliterans (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Vasculitis (Vascular disorders) | 1 | 1
Aneurysm (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Hypoperfusion (Vascular disorders) | 1 | 0
Iliac vein occlusion (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 1 | 0
Thrombosed varicose vein (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Wound haemorrhage (Vascular disorders) | 1 | 0
Haemorrhagic infarction (Vascular disorders) | 0 | 2
Aneurysm arteriovenous (Vascular disorders) | 0 | 1
Aortic rupture (Vascular disorders) | 0 | 1
Arterial disorder (Vascular disorders) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 15 | 12
Gout (Metabolism and nutrition disorders) | 9 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2
Cachexia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Haemosiderosis (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Neuroglycopenia (Metabolism and nutrition disorders) | 0 | 1
Underweight (Metabolism and nutrition disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 24 | 21
Prostatitis (Reproductive system and breast disorders) | 5 | 3
Uterine polyp (Reproductive system and breast disorders) | 2 | 2
Prostatomegaly (Reproductive system and breast disorders) | 1 | 2
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Prostatism (Reproductive system and breast disorders) | 1 | 1
Colpocele (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0
Genital prolapse (Reproductive system and breast disorders) | 1 | 0
Uterine cervical erosion (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Breast haematoma (Reproductive system and breast disorders) | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Peyronie's disease (Reproductive system and breast disorders) | 0 | 1
Prostatic disorder (Reproductive system and breast disorders) | 0 | 1
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1
Spermatocele (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Varicocele (Reproductive system and breast disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 17 | 12
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 2
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Chest pain (General disorders) | 9 | 6
General physical health deterioration (General disorders) | 4 | 3
Non-cardiac chest pain (General disorders) | 3 | 7
Asthenia (General disorders) | 3 | 2
Hernia obstructive (General disorders) | 3 | 0
Pyrexia (General disorders) | 2 | 6
Multi-organ failure (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 1 | 3
Gait disturbance (General disorders) | 1 | 2
Hernia (General disorders) | 1 | 2
Generalised oedema (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Catheter site pain (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Implant site effusion (General disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Pain (General disorders) | 0 | 2
Catheter thrombosis (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Fat tissue increased (General disorders) | 0 | 1
Hyperplasia (General disorders) | 0 | 1
Hypertrophy (General disorders) | 0 | 1
Perforated ulcer (General disorders) | 0 | 1
Puncture site haemorrhage (General disorders) | 0 | 1
Cataract (Eye disorders) | 17 | 18
Glaucoma (Eye disorders) | 2 | 3
Eye haemorrhage (Eye disorders) | 2 | 2
Retinal vein thrombosis (Eye disorders) | 2 | 0
Vitreous haemorrhage (Eye disorders) | 2 | 0
Retinal detachment (Eye disorders) | 1 | 6
Retinal haemorrhage (Eye disorders) | 1 | 1
Diplopia (Eye disorders) | 1 | 0
Episcleritis (Eye disorders) | 1 | 0
Pupils unequal (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Retinal disorder (Eye disorders) | 1 | 0
Retinal vascular thrombosis (Eye disorders) | 1 | 0
Retinoschisis (Eye disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 2
Optic ischaemic neuropathy (Eye disorders) | 0 | 2
Eye disorder (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Depression (Psychiatric disorders) | 4 | 6
Confusional state (Psychiatric disorders) | 4 | 4
Completed suicide (Psychiatric disorders) | 3 | 3
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 3
Psychotic disorder (Psychiatric disorders) | 1 | 2
Alcohol abuse (Psychiatric disorders) | 1 | 1
Stress (Psychiatric disorders) | 1 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 1 | 0
Delusional disorder, persecutory type (Psychiatric disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Somatisation disorder (Psychiatric disorders) | 1 | 0
Delusional disorder, unspecified type (Psychiatric disorders) | 0 | 1
Depressive symptom (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1
Neurosis (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Acanthosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 8 | 10
Goitre (Endocrine disorders) | 3 | 3
Toxic nodular goitre (Endocrine disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Hyperaldosteronism (Endocrine disorders) | 1 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 8 | 9
Sudden hearing loss (Ear and labyrinth disorders) | 2 | 0
Vestibular disorder (Ear and labyrinth disorders) | 2 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 2
Hearing impaired (Ear and labyrinth disorders) | 1 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 1
Vertigo labyrinthine (Ear and labyrinth disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Sick sinus syndrome (Cardiac disorders) | 2 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac amyloidosis (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac perforation (Cardiac disorders) | 0 | 1
Dressler's syndrome (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Sinoatrial block (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 5 | 1
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 2 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 4
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 1 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0
Muscular dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 | 1
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Colon operation (Surgical and medical procedures) | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Retinal operation (Surgical and medical procedures) | 1 | 0
Wound drainage (Surgical and medical procedures) | 1 | 0
Alcohol detoxification (Surgical and medical procedures) | 0 | 1
Dacryocystorhinostomy (Surgical and medical procedures) | 0 | 1
Eventration procedure (Surgical and medical procedures) | 0 | 1
Intestinal stoma (Surgical and medical procedures) | 0 | 1
Intraocular lens repositioning (Surgical and medical procedures) | 0 | 1
Renal cyst excision (Surgical and medical procedures) | 0 | 1
International normalised ratio increased (Investigations) | 2 | 5
Haemoglobin decreased (Investigations) | 1 | 3
Weight decreased (Investigations) | 1 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Aspiration bronchial (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 2
Drug hypersensitivity (Immune system disorders) | 1 | 1
Allergy to arthropod sting (Immune system disorders) | 1 | 0
Bedridden (Social circumstances) | 0 | 1
Elderly (Social circumstances) | 0 | 1
Social stay hospitalisation (Social circumstances) | 0 | 1
Walking disability (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Irbesartan (N=4518) | Placebo (N=4498)
Any infections and infestations (Infections and infestations) | 1369 | 1369
Bronchitis (Infections and infestations) | 255 | 251
Nasopharyngitis (Infections and infestations) | 225 | 238
Any nervous system disorders (Nervous system disorders) | 1067 | 917
Dizziness (Nervous system disorders) | 529 | 399
Any gastrointestinal disorders (Gastrointestinal disorders) | 1044 | 1059
Any musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 884 | 930
Any general disorders and administration site conditions (General disorders) | 836 | 858
Oedema peripheral (General disorders) | 259 | 302
Any vascular disorders (Vascular disorders) | 784 | 686
Hypotension (Vascular disorders) | 350 | 193
Hypertension (Vascular disorders) | 209 | 273
Any respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 772 | 782
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 333 | 330
Any injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 569 | 582
Any skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 464 | 465
Any cardiac disorders (Cardiac disorders) | 444 | 455
Any metabolism and nutrition disorders (Metabolism and nutrition disorders) | 383 | 384
Any eye disorders (Eye disorders) | 345 | 336
Any renal and urinary disorders (Renal and urinary disorders) | 344 | 282
Any neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 296 | 358
Any investigations (Investigations) | 276 | 297
Any psychiatric disorders (Psychiatric disorders) | 260 | 275

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the study will be made jointly in the name of all wholehearted collaborators. Other papers will be authored based on the contributions of the individuals to the overall study. Substudies with scientific merit which have received prior approval from the Steering Committee (SC) may be published in the names of the contributing investigators. A copy of all manuscripts will be provided to the sponsors for their review. The final decision to publish articles will be made by the SC.